CLINICAL TRIAL: NCT04111809
Title: Assessment of 4 Bone Turnover Markers (C-terminal Telopeptides of Type I Collagene (CTX), Amino-terminal Telopeptide of Type 1 Collagen (NTX), Dickkopf-1 (DKK-1) and Sclerostin (SOST)) in Multiple Myeloma Patients Treated With Intravenous Bisphosphonate
Brief Title: Study of 4 Bone Turnover Markers in Patients With Multiple Myeloma Treated With Intravenous Bisphosphonate in Routine Care
Acronym: AMBROBiMM
Status: Terminated | Type: Observational
Why Stopped: Inability to conduct the study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Intergroupe Francophone du Myelome (Network); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APH190198
Record Dates: First submitted 2019-09-04; First posted 2019-10-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; intravenous bisphosphonate; bone markers
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum plasma urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- intravenous biphosphonate: Patients treated with intravenous bisphosphonate until 12 months in routine care
  Interventions: Biological: Blood and urine collection

INTERVENTIONS:
Biological: Blood and urine collection — collected 10 mL of blood and 15 mL of urine every 2 months until 12 months

SUMMARY:
The aim of this study is looking at the Kinetics of bone turnover markers (C-terminal telopeptides of type I collagene (CTX), amino-terminal telopeptide of type 1 collagen (NTX), Dickkopf-1 (DKK-1) and Sclerostin (SOST)) in serum and urine until 12 months in Patients with Multiple Myeloma Treated With intravenous bisphosphonates in routine care.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 65 to 75 years of age
2. Patient with symptomatic multiple myeloma as defined by the criteria of the IMWG
3. Need to introduced an antiresorptive bone treatment by intravenous bisphosphonate with bone imaging mapping (PET-scanner preferentially) in routine care
4. Ability and willingness to follow scheduled visits with requested biological samples

Exclusion Criteria

- Patients previously treated with intravenous biphosphonate

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: no description
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Changes in bone turnover markers | Baseline, then every 2 months in 12 months
  bone turnover markers include: C-terminal telopeptides of type I collagene (CTX) in serum, amino-terminal telopeptide of type 1 collagen (NTX) in urine, Dickkopf-1 (DKK-1) and Sclerostin (SOST) in plasma

SECONDARY OUTCOMES:
time to maximum variation of bone turnover markers | Baseline, then every 2 months in 12 months
  CTX, NTX, DKK-1 and SOST
Doses of intravenous bisphosphonate | Up to 12 months
  To study the relationship between doses and bone turnover markers
Rate of intravenous bisphosphonate | Up to 12 months
  To study the relationship between doses and bone turnover markers
evolution of bone lesions by imaging | Up to 12 months
  evolution of bone lesions by imaging
Number of new bone events | Up to 12 months
Number of adverse events likely to be related to bisphosphonate | Up to 12 months
Changes in Monoclonal protein | Baseline, then every 2 months in 12 months
  To evaluated response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Necker Hospital, Adult haematology department, Paris, France

IPD SHARING:
Plan to Share IPD: No